CLINICAL TRIAL: NCT06082232
Title: Intrathecal Dexmedetomidine Versus Midazolam as Adjuvants With Intrathecal Bupivacaine for Postoperative Analgesia in High Tibial Osteotomy. A Randomized, Prospective, Double- Blinded, Comparative Study.
Brief Title: Adjuvants With Intrathecal Bupivacaine for Postoperative Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Sayed Ali Farghali, Doctor, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Postoperative analgesia in HTO
Record Dates: First submitted 2023-10-04; First posted 2023-10-13 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Midazolam; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group M (midazolam group) (Active Comparator): includes thirty patients who receive intrathecal 4 mL (20 mg) 0.5% hyperbaric bupivacaine and 1 mg midazolam (8 units of 5 mg/mL preservative-free midazolam loaded in a 40 unit insulin syringe).
  Interventions: Drug: Midazolam; Drug: Bupivacain
- Group D(dexmedetomidine group) (Active Comparator): includes thirty patients who receive intrathecal 4 mL (20 mg) 0.5% hyperbaric bupivacaine and 5 mcg dexmedetomidine (2 units of 100 mcg/mL preservative-free dexmedetomidine loaded in a 40 unit insulin syringe).
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacain
- Group C(control group) (Placebo Comparator): includes thirty patients who receive intrathecal 4 mL (20 mg) 0.5% hyperbaric bupivacaine and 0.5 mL of 0.9% saline .
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Dexmedetomidine — Under strict aseptic conditions, a lumbar puncture will be performed with selective technique in sitting position at L2-3 or L3-4 interspaces with midline approach using a 25-G Quincke's needle. After achieving the free flow of cerebrospinal fluid, the study drug will be injected into the subarachnoid space, immediately after injection the patient will be asked for supine position.
  Arms: Group D(dexmedetomidine group)
Drug: Midazolam — 1 mg midazolam intrathecal administration
  Arms: Group M (midazolam group)
Drug: Bupivacain — 20 mg bupivacaine intrathecal administration

SUMMARY:
The aim of this study is to compare the postoperative analgesic effect of intrathecal dexmedetomidine combined with bupivacaine and midazolam combined with bupivacaine in high tibial osteotomy.

DETAILED DESCRIPTION:
With more than 80% of patients experiencing acute pain following surgical procedures, and half of them reporting inadequate pain therapy, the control and management of post-surgical pain remains one of the most challenging aims of modern anesthesia.

Adequate postoperative pain control is an important part of postoperative care treatment. World Health Organization, as well as International Association for the Study of Pain, have emphasized its significance for patients well-being, and determined pain relief to be a human right and the occurrence of pain as fifth vital sign.

Local anesthetic, bupivacaine, is the most common agent used for spinal anesthesia but has relatively short duration of action. Many adjuvants to local anesthetics have been used intrathecally to improve the quality of intraoperative analgesia and prolong it in the postoperative period.

Diverse classes of drugs such as opioids , epinephrine , neostigmine , magnesium , midazolam , ketamine , and clonidine have been added to intrathecal local anaesthetics in an attempt to prolong analgesia and reduce the incidence of adverse events.

Opioids are commonly added to local anaesthetics to produce spinal and epidural anesthesia. However, significant adverse effects such as, urinary retention, respiratory depression, hemodynamic instability, pruritus and occasionally severe nausea and vomiting, may limit their use .

α2-adrenergic agonists are new neuraxial adjuvants being studied to improve the quality of subarachnoid blockade regarding both sensory and motor blockades. There are many studies supporting their efficacy as adjuvants individually.

Dexmedetomidine, a highly specific, potent, and selective α2-adrenergic agonist, provides stable hemodynamic conditions and good quality of intraoperative and prolonged postoperative analgesia with minimal side effects.

Discovery of benzodiazepine receptors in spinal cord in 1977 triggered the use of intrathecal midazolam for prolongation of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years.
* Gender: Both males and females.
* Scheduled patients for High tibial osteotomy under spinal anesthesia.
* American Society of Anesthesiologists (ASA) physical status: I and II

Exclusion Criteria:

* Patient refusal
* Allergy to the studied drugs.
* Patients with contraindications to spinal anesthesia.
* Patients with advanced decompensated cardiac, respiratory,renal or hepatic diseases
* Coagulopathy or thrombocytopenia
* CNS diseases as epilepsy, stroke or psychiatric illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to first analgesic request | 24 hours
  Time to first analgesic request calculated from the administration of local anesthetic

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  Total analgesic consumption in the first 24 hour .
Incidence of complications | 24 hours
  Incidence of complications (bradycardia , hypotension ,nausea and vomiting).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Youssef, Study Chair — Assiut University; Mahmoud Kamel, Study Director — Assiut University

REFERENCES:
- [Background] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977
- [Background] Chaney MA. Side effects of intrathecal and epidural opioids. Can J Anaesth. 1995 Oct;42(10):891-903. doi: 10.1007/BF03011037. PMID 8706199
- [Background] Kanazi GE, Aouad MT, Jabbour-Khoury SI, Al Jazzar MD, Alameddine MM, Al-Yaman R, Bulbul M, Baraka AS. Effect of low-dose dexmedetomidine or clonidine on the characteristics of bupivacaine spinal block. Acta Anaesthesiol Scand. 2006 Feb;50(2):222-7. doi: 10.1111/j.1399-6576.2006.00919.x. PMID 16430546
- [Background] Mohler H, Okada T. Benzodiazepine receptor: demonstration in the central nervous system. Science. 1977 Nov 25;198(4319):849-51. doi: 10.1126/science.918669.